CLINICAL TRIAL: NCT02977052
Title: Multicenter Phase 2 Study to Identify of the Optimal Neo-Adjuvant Combination Scheme of Ipilimumab and Nivolumab (OpACIN-neo)
Brief Title: Optimal Neo-adjuvant Combination Scheme of Ipilimumab and Nivolumab
Acronym: OpACIN-neo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16OPN; 2016-001984-35 (EudraCT Number); CA209-701 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2016-11-21; First posted 2016-11-30 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Malignant Melanoma Stage III
Keywords: Melanoma; Ipilimumab; Nivolumab; Neo-adjuvant
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab; Surgical Procedures, Operative; Blood Specimen Collection; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A: 2 courses ipi 3 + nivo 1 (Experimental): Patients receive 2 courses standard combination of ipilimumab 3 mg/kg + nivolumab 1 mg/kg q3wk prior to surgery at week 6. Blood for PBMCs and biopsies will be taken for translation research.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Procedure: Surgery; Procedure: Blood for PBMCs; Procedure: Biopsies
- Arm B: 2 courses ipi 1 + nivo 3 (Experimental): Patients receive 2 courses ipilimumab 1 mg/kg + nivolumab 3 mg/kg q3wk prior to surgery at week 6. Blood for PBMCs and biopsies will be taken for translation research.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Procedure: Surgery; Procedure: Blood for PBMCs; Procedure: Biopsies
- Arm C: 2 courses ipi 3 + 2 courses nivo 3 (Experimental): Patients receive 2 courses of ipilimumab 3 mg/kg q3wks, directly followed (> 2 hours and < 24 hours) by 2 courses nivolumab 3 mg/kg every 2 weeks prior to surgery at week 6. Blood for PBMCs and biopsies will be taken for translation research.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Procedure: Surgery; Procedure: Blood for PBMCs; Procedure: Biopsies
- PRADO extension cohort (Experimental): Patients will be treated with 2 courses ipilimumab and nivolumab at the dose level defined as the winner dosing scheme from OpACIN-neo, which is the dosing schedule of arm B.
  Surgery and adjuvant therapy
  * Patients achieving a pCR or pnCR will not undergo CLND and will not receive any adjuvant treatment. Structural follow-up will be perfomed every 12 weeks by CT, ultrasound of regional lymph nodes.
  * Patients achieving a pPR will undergo CLND and start structural follow-up (including CT and physical examination) every 12 weeks thereafter without any adjuvant treatment.
  * Patients achieving no response (pNR) will undergo CLND and start at week 12 with adjuvant nivolumab 480mg q4wks for 52 weeks + radiotherapy (according to patient's and physicians' decision). In patients that are BRAF V600E/K mutation positive, adjuvant BRAF+MEK
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Procedure: Surgery; Procedure: Blood for PBMCs; Procedure: Biopsies

INTERVENTIONS:
Drug: Ipilimumab
Drug: Nivolumab
Procedure: Surgery — Surgery will be done at 6 weeks
Procedure: Blood for PBMCs — Blood will be taken for translational research on PBMCs
Procedure: Biopsies — Biopsies will be taken during screening and at relapse.

SUMMARY:
This is an open-label three-arm phase 2 trial (including a Simon stage 2 design) consisting of 90 stage III melanoma patients randomized 1:1:1 to receive either 2 courses 3 mg/kg ipilimumab + 1 mg/kg nivolumab every 3 weeks (Arm A), 2 courses 1 mg/kg ipilimumab + 3 mg/kg nivolumab every 3 weeks (Arm B), or 2 courses ipilimumab 3 mg/kg, directly followed by 2 courses nivolumab 3 mg/kg every 2 weeks (Arm C). All three treatment arms are applied prior to surgery at week 6, 30 patients per arm. Patients will be stratified according to treatment center. An interim analysis will be performed after 13 patients have been included in each arm, thus in total 39 patients have been included.

PRADO extension cohort The trial will enroll in total about 100-110 melanoma patients with macroscopic stage III disease (RECIST measurable disease); inclusion will stop when 50 patients have achieved a pCR or pnCR. All patients will be treated (after marker placement into the largest lymph node metastasis) with the winner combination identified in the first part of the OpACIN-neo study which is 2 courses ipilimumab 1mg/kg + nivolumab 3mg/kg, q3wks. After 6 weeks of treatment, the patients will undergo only surgical resection of the marked index lymph node. Thereafter subsequent surgery and adjuvant therapy will be performed according to the achieved pathologic response.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* World Health Organization (WHO) Performance Status 0 or 1
* Cytologically or histologically confirmed resectable stage III melanoma with one or more macroscopic lymph node metastases (measurable according to RECIST 1.1), that can be biopsied, and no history of in-transit metastases within the last 6 months
* No other malignancies, except adequately treated and a cancer-related life-expectancy of more than 5 years
* Patient willing to undergo triple tumor biopsies and extra blood withdrawal during screening and in case of relapse
* No prior immunotherapy targeting CTLA-4, PD-1 or PD-L1
* No immunosuppressive medications within 6 months prior study inclusion
* Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Neutrophils ≥1.5x109/L, Platelets ≥100 x109/L, Hemoglobin ≥5.5 mmol/L, Creatinine ≤1.5x ULN, AST ≤ 1.5 x ULN, ALT ≤ 1.5 x ULN, Bilirubin ≤1.5 X ULN
* Normal LDH
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contra-ception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of ipilimumab + nivolumab
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product
* Women who are not of childbearing potential (i.e., who are postmenopausal), or surgically sterile as well as azoospermic men do not require contraception
* Patient is capable of understanding and complying with the protocol requirements and has signed the Informed Consent document.

Exclusion Criteria:

* Distantly metastasized melanoma
* History of in-transit metastases within the last 6 months
* No measurable lesion according to RECIST 1.1
* Subjects with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for subjects with vitiligo or resolved childhood asthma/atopy
* Prior CTLA-4 or PD-1/PD-L1 targeting immunotherapy
* Radiotherapy prior or post-surgery
* Patients will be excluded if they test positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody), indicating acute or chronic infection
* Patients will be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Allergies and Adverse Drug Reaction

  * History of allergy to study drug components
  * History of severe hypersensitivity reaction to any monoclonal antibody
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events;
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids;
* Use of other investigational drugs before study drug administration 30 days and 5 half-times before study inclusion
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2016-11-24 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by the frequency of grade 3/4 immune-related adverse events, using CTCAE 4.03 | During the first 12 weeks.
Response rate according to RECIST 1.1 | At 6 weeks
Pathological response according to central pathological revision, according to pathological response criteria | At 6 weeks
Pathologic response rate according to central revision of the marked index lymph node | At 6 weeks, prior surgery
RFS at 24 months in patients achieving pCR or pnCR in their marked index lymph node and did not undergo CLND. RFS will be calculated from date of resection of the marked lymph node. | 24 months
RFS at 24 months in patients with pNR and being subsequently treated with adjuvant nivolumab+optional radiotherapy (or dabrafenib/trametinib if BRAFV600E pos. and treatment is approved). RFS will be calculated from day of resection of marked lymph node. | 24 months

SECONDARY OUTCOMES:
Recurrence Free Survival | 3 years after treatment initiation
Description of late adverse events using CTCAE 4.03 | Up to 3 years after treatment initiation until new treatment
Description of associations of mutational load, RNA tumor signatures, and tumor educated platelet signatures with tumor immune infiltrates and response | At 6 weeks
Response rate according to RECIST 1.1 at week 6 | At 6 weeks
RFS at 2, 3 and 5 years | Up to 5 years after treatment

OTHER OUTCOMES:
EFS at 2, 3 and 5 years | Up to 5 years after treatment
DMFS at 2, 3 and 5 years | Up to 5 years after treatment
OS at 2, 3 and 5 years | Up to 5 years after treatment
Grade 3/4 immune-related adverse event rate according to CTCAE v4.03 within the first 12 weeks | At 12 weeks
• Surgical complication rates according to Clavien-Dindo surgical classification of only marked index lymph node resection vs. CLND | At 12 weeks
• Description of late adverse event (up to 3 years after treatment initiation) according to CTCAE v4.03 | Up to 3 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christian Blank, Prof., Study Chair — Medical oncologist/researcher
Locations (4):
- Melanoma Institute Australia, Sydney, New South Wales, Australia
- Medical University of Vienna, Vienna, Austria
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoeijmakers LL, Dimitriadis P, Wijnen SCMA, Reijers ILM, Lopez-Yurda M, Menzies AM, Broeks A, Cornelissen S, Torres Acosta A, van der Wal A, Saw RPM, Versluis JM, van Houdt WJ, Wouters MW, Romano J, Rozeman EA, Grijpink-Ongering LG, Kapiteijn E, van der Veldt AAM, Suijkerbuijk KPM, Eriksson H, Hospers GAP, van der Hage JA, Grunhagen DJ, Witkamp AJ, Lijnsvelt JM, Klop WMC, Zuur CL, Bruining A, Al-Mamgani A, Pennington TE, Shannon KF, Ch'ng S, Colebatch AJ, Gonzalez M, Spillane AJ, Haanen JBAG, Rawson RV, Scolyer RA, van de Wiel BA, van Akkooi ACJ, Long GV, Blank CU. Neoadjuvant ipilimumab plus nivolumab in melanoma: 5-year survival and biomarker analysis from the phase 2 PRADO-trial. Nat Med. 2026 Jan 28. doi: 10.1038/s41591-025-04158-9. Online ahead of print. PMID 41606118
- [Derived] Fraterman I, Reijers ILM, Dimitriadis P, Broeks A, Gonzalez M, Menzies AMM, Lopez-Yurda M, Kapiteijn E, van der Veldt AAM, Suijkerbuijk KPM, Hospers GAP, Long GV, Blank CU, van de Poll-Franse LV. Association between pretreatment emotional distress and neoadjuvant immune checkpoint blockade response in melanoma. Nat Med. 2023 Dec;29(12):3090-3099. doi: 10.1038/s41591-023-02631-x. Epub 2023 Nov 13. PMID 37957378
- [Derived] Hoefsmit EP, Vollmy F, Rozeman EA, Reijers ILM, Versluis JM, Hoekman L, van Akkooi ACJ, Long GV, Schadendorf D, Dummer R, Altelaar M, Blank CU. Systemic LRG1 Expression in Melanoma is Associated with Disease Progression and Recurrence. Cancer Res Commun. 2023 Apr 20;3(4):672-683. doi: 10.1158/2767-9764.CRC-23-0015. eCollection 2023 Apr. PMID 37089863
- [Derived] Zijlker LP, van der Burg SJC, Blank CU, Zuur CL, Klop WMC, Wouters MWMJ, van Houdt WJ, van Akkooi ACJ. Surgical outcomes of lymph node dissections for stage III melanoma after neoadjuvant systemic therapy are not inferior to upfront surgery. Eur J Cancer. 2023 May;185:131-138. doi: 10.1016/j.ejca.2023.03.003. Epub 2023 Mar 7. PMID 36989829
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215
- [Derived] Reijers ILM, Menzies AM, van Akkooi ACJ, Versluis JM, van den Heuvel NMJ, Saw RPM, Pennington TE, Kapiteijn E, van der Veldt AAM, Suijkerbuijk KPM, Hospers GAP, Rozeman EA, Klop WMC, van Houdt WJ, Sikorska K, van der Hage JA, Grunhagen DJ, Wouters MW, Witkamp AJ, Zuur CL, Lijnsvelt JM, Torres Acosta A, Grijpink-Ongering LG, Gonzalez M, Jozwiak K, Bierman C, Shannon KF, Ch'ng S, Colebatch AJ, Spillane AJ, Haanen JBAG, Rawson RV, van de Wiel BA, van de Poll-Franse LV, Scolyer RA, Boekhout AH, Long GV, Blank CU. Personalized response-directed surgery and adjuvant therapy after neoadjuvant ipilimumab and nivolumab in high-risk stage III melanoma: the PRADO trial. Nat Med. 2022 Jun;28(6):1178-1188. doi: 10.1038/s41591-022-01851-x. Epub 2022 Jun 5. PMID 35661157
- [Derived] Versluis JM, Reijers ILM, Rozeman EA, Menzies AM, van Akkooi ACJ, Wouters MW, Ch'ng S, Saw RPM, Scolyer RA, van de Wiel BA, Schilling B, Long GV, Blank CU. Neoadjuvant ipilimumab plus nivolumab in synchronous clinical stage III melanoma. Eur J Cancer. 2021 May;148:51-57. doi: 10.1016/j.ejca.2021.02.012. Epub 2021 Mar 15. PMID 33735809
- [Derived] Rozeman EA, Hoefsmit EP, Reijers ILM, Saw RPM, Versluis JM, Krijgsman O, Dimitriadis P, Sikorska K, van de Wiel BA, Eriksson H, Gonzalez M, Torres Acosta A, Grijpink-Ongering LG, Shannon K, Haanen JBAG, Stretch J, Ch'ng S, Nieweg OE, Mallo HA, Adriaansz S, Kerkhoven RM, Cornelissen S, Broeks A, Klop WMC, Zuur CL, van Houdt WJ, Peeper DS, Spillane AJ, van Akkooi ACJ, Scolyer RA, Schumacher TNM, Menzies AM, Long GV, Blank CU. Survival and biomarker analyses from the OpACIN-neo and OpACIN neoadjuvant immunotherapy trials in stage III melanoma. Nat Med. 2021 Feb;27(2):256-263. doi: 10.1038/s41591-020-01211-7. Epub 2021 Feb 8. PMID 33558721
- [Derived] Rozeman EA, Menzies AM, van Akkooi ACJ, Adhikari C, Bierman C, van de Wiel BA, Scolyer RA, Krijgsman O, Sikorska K, Eriksson H, Broeks A, van Thienen JV, Guminski AD, Acosta AT, Ter Meulen S, Koenen AM, Bosch LJW, Shannon K, Pronk LM, Gonzalez M, Ch'ng S, Grijpink-Ongering LG, Stretch J, Heijmink S, van Tinteren H, Haanen JBAG, Nieweg OE, Klop WMC, Zuur CL, Saw RPM, van Houdt WJ, Peeper DS, Spillane AJ, Hansson J, Schumacher TN, Long GV, Blank CU. Identification of the optimal combination dosing schedule of neoadjuvant ipilimumab plus nivolumab in macroscopic stage III melanoma (OpACIN-neo): a multicentre, phase 2, randomised, controlled trial. Lancet Oncol. 2019 Jul;20(7):948-960. doi: 10.1016/S1470-2045(19)30151-2. Epub 2019 May 31. PMID 31160251